CLINICAL TRIAL: NCT02875821
Title: Effects of Ipragliflozin on Excessive Fat in Type 2 Diabetes Patients With Non-alcoholic Fatty Liver Disease Treated With Metformin and Pioglitazone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-1115
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes With Non-alcoholic Fatty Liver (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ipragliflozin; Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group IMP (Experimental): Group IMP (Ipragliflozin with Metformin with Pioglitazone)
  Interventions: Drug: Ipragliflozin
- Group MP (Active Comparator): Group MP (Metformin with Pioglitazone)
  Interventions: Drug: metformin with pioglitazone

INTERVENTIONS:
Drug: Ipragliflozin — Patients treated with ipragliflozin (50 mg/day) as add on therapy to metformin and pioglitazone dual therapy (triple therapy) for 6 months. During whole periods of study, subjects are educated for nutrition and exercise. (Experimental Group)
  Other Names: Suglat®
  Arms: Group IMP
Drug: metformin with pioglitazone — Patients maintain metformin and pioglitazone dual therapy for 6 months. During whole periods of study, subjects are educated for nutrition and exercise. (Control group)
  Arms: Group MP

SUMMARY:
In this study, the investigators investigate beneficial effects of ipragliflozin, newly developted SGLT2 inhibitor, on reduction in visceral fat area and degree of fatty liver in subjects with T2DM when added to metformin and pioglitazone therapy.

DETAILED DESCRIPTION:
Pioglitazone, a peroxisome proliferator-activated receptor-γ (PPARγ) agonist increase insulin sensitivity in peripheral tissue and liver by protecting non-adipose tissues against excessive lipid overload and by balancing the secretion of adipocytokines.

However, PPARγ is a key transcription factor that induces the differentiation adipocyte maturation and stimulates the induction of enzymes involved in lipogenesis. As a result, the effect of pioglitazone is generally accompanied by weight gain and an increase in amount of subcutaneous fat.

Obesity would coexist with fatty liver disease and both conditions aggravate hyperglycemia in diabetes. According to recent study, up-regulated PPARγ expression in liver was reported in obesity with hepatic steatosis which implies pioglitazone might induce fatty liver disease.

A novel oral antidiabetic drug, sodium glucose cotransporter 2 (SGLT2) inhibitor reduces renal glucose reabsorption and increasing renal glucose excretion thereby promoting energy loss. As a result, it prevents weight gain and fluid retention which might counteract the unfavorable effects of pioglitazone treatment.

No study has been conducted on the additional effect on obesity and fatty liver of ipragliflozin in T2DM patients treated with pioglitazone and metformin.

In this study, the investigators investigate beneficial effects of ipragliflozin, newly developted SGLT2 inhibitor, on reduction in visceral fat area and degree of fatty liver in subjects with T2DM when added to metformin and pioglitazone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Diagnosed as NAFLD
* Age of 20~75
* On metformin + pioglitazone treatment with stable dose for at least 8 weeks
* Adequate glycemic control: HbA1c ≤ 9.5%
* Overweight & obese: BMI ≥ 23 kg/m2
* Subject is male, or subject is female who is highly unlikely to conceive
* Understands the study procedure, alternatives, and risks and voluntarily agrees to participate by giving written informed consent

Exclusion Criteria:

* Type 1 diabetes, Secondary diabetes, gestational diabetes
* Heavy alcoholics (men ≥210 g of alcohol per week, women ≥140 g of alcohol per week)
* Underlying chronic liver disease (hemochromatosis, liver cell carcinoma, autoimmune liver disease, liver cirrhosis, chronic viral hepatitis [except hepatitis B carrier], Wilson's disease)
* Patients on medication causes hepatic steatosis (e.g.amiodarone, methotrexate, tamoxifen, valproate, corticosteroids, etc)
* Allergy or hypersensitivity to target medication or any of its components
* Renal failure, moderate or severe renal impairment (estimated glomerular filtration rate < 60 mL/min/1.73 m2), or ongoing dialysis
* Abnormal liver function (AST/ALT > x10 upper normal limit)
* On taking weight loss medication
* History of alcohol or drug abuse in the previous 3 months
* Premenopausal women who are nursing or pregnant
* Human immunodeficiency virus (HIV) or human immunodeficiency virus (AIDS)
* Diabetic ketoacidosis
* Severe infection, severe trauma

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
changes in visceral fat area | 6 months
  The visceral fat area is measured by dual-energy x-ray absorptiometry (DEXA) at baseline and after 6 months treatment

SECONDARY OUTCOMES:
Changes in subcutaneous fat area | 6 months after treatment
  The subcutaneous fat area is measured by dual-energy x-ray absorptiometry (DEXA) and fat computed tomography (CT) at baseline and after 6 months treatment.
Changes in liver fat | 6 months after treatment
  Changes in the degree of fatty liver is measured by fibroscan using controlled attenuation parameter (CAP) score.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided